CLINICAL TRIAL: NCT03448978
Title: Phase I Safety and Feasibility Study of Autologous CD8+ T-cells Transiently Expressing a Chimeric Antigen Receptor Directed to B-Cell Maturation Antigen in Patients With Multiple Myeloma
Brief Title: Autologous CD8+ T-cells Expressing an Anti-BCMA CAR in Patients With Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase 1 enrollment completed. Further clinical development terminated
Sponsor: Cartesian Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 241-59-88
Record Dates: First submitted 2018-01-24; First posted 2018-02-28 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma
Keywords: Descartes-08; CAR T Cell; CART; CAR-T; CAR T-Cell; Multiple Myeloma; BCMA; B-cell maturation antigen; B cell maturation antigen
MeSH Terms: conditions — Multiple Myeloma | interventions — Immunotherapy, Adoptive; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Descartes-08 plus fludarabine/cyclophosphamide pretreat (Experimental): Autologous CD8+ T-cells transiently expressing an anti-BCMA chimeric antigen receptor
  Interventions: Biological: Descartes-08; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Descartes-08 — autologous CD8+ T-cells transiently expressing an anti-BCMA chimeric antigen receptor
  Other Names: CAR-T cells
Drug: Fludarabine — intravenous fludarabine
Drug: Cyclophosphamide — intravenous cyclophosphamide

SUMMARY:
This Phase I study will test the safety and anti-myeloma activity of ascending doses of Descartes-08 (autologous CD8+ T-cells expressing an anti-BCMA chimeric antigen receptor) in eligible patients with active multiple myeloma.

ELIGIBILITY:
Inclusion Criteria (condensed):

* Multiple myeloma that is double-refractory to a proteasome inhibitor (PI) and an immunomodulatory drug (IMiD) after at least 2 prior lines of therapy OR have failed at least 3 prior lines of therapy
* Measurable disease activity as indicated by serum or urine M-protein, serum free light chain, biopsy-proven plasmacytoma, >5% bone marrow plasma cells.
* Adequate vital organ function as indicated by ANC (>1000/uL), platelet count (>50,000/uL), hemoglobin (>8 g/dL), serum ALT and AST (each <3.0 x upper limit of normal), total bilirubin (<2 mg/dL), creatinine clearance (>30 mL/min), and cardiac ejection fraction (>45%)

Exclusion Criteria (condensed):

NOTE: Prior anti-BCMA or CAR-T therapy is NOT exclusionary

* Active plasma cell leukemia
* Pregnant or lactating
* Active, uncontrolled infection
* Active and severe auto-immune disease
* Active arrhythmia, or obstructive or restrictive pulmonary disease
* Central nervous system disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Incidence (number) of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 weeks
  Incidence (number) of Treatment-Emergent Adverse Events [Safety and Tolerability]. Descriptive statistics by incidence rate, body system classification, severity, and causality [per protocol definitions]

SECONDARY OUTCOMES:
Treatment response | 1, 3, 6, 9 and 12 months
  IMWG treatment response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Metin Kurtoglu, MD, PhD, Study Director — Cartesian Therapeutics
Locations (3):
- United States (3):
  - The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Virgina Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No